CLINICAL TRIAL: NCT02838680
Title: Transfemoral Replacement of Aortic Valve With HLT MeriDIAN Valve Feasibility Trial CANADA
Acronym: RADIANT CANADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLT1502
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic stenosis; transcatheter aortic valve replacement (TAVR)
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HLT Transcatheter Aortic Valve System (Experimental): Transcatheter aortic valve replacement with HLT Transcatheter Aortic Valve System
  Interventions: Device: HLT Transcatheter Aortic Valve System

INTERVENTIONS:
Device: HLT Transcatheter Aortic Valve System — Transcatheter aortic valve replacement with HLT Transcatheter Aortic Valve System

SUMMARY:
To evaluate the safety and performance of the HLT System in patients with severe aortic stenosis who present at high risk for aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 70 years of age or older
2. Echocardiographic or hemodynamic based evidence of calcific (senile) aortic stenosis with one of the following: aortic valve EOA <1.0 cm2 or 0.6 cm2/m2 , mean aortic valve gradient >40 mmHg or peak aortic valve velocity >4 m/sec
3. Symptomatology due to aortic stenosis resulting in one of the following:

   1. NYHA Functional Classification of II or greater
   2. Presence of angina
   3. Presence of syncope
4. Aortic valve annular diameter ≥ 24 and ≤26 mm measured by MSCT based on area or perimeter
5. STS score of ≥8, or documented heart team agreement of high risk for surgical aortic valve replacement (SAVR) due to frailty or comorbidities.
6. Geographically available, willing to comply with follow up and able to provide written informed consent

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve, or noncalcified aortic valve; or valve eccentricity (calcific or otherwise) that in the opinion of the investigator could compromise procedural success.
2. Patients at high risk for coronary obstruction in the opinion of the investigator (e.g. combination of a coronary height < 12 mm and coronary sinus diameter < 30 mm)
3. Patients with low flow/low gradient aortic stenosis
4. Patients with significant annular calcification (e.g. Agatston score > 4000)
5. Pre-existing prosthetic heart valve in any position, or prosthetic ring
6. Severe aortic, mitral or tricuspid valve regurgitation
7. Moderate to severe mitral stenosis
8. Myocardial infarction within the past 30 days*
9. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
10. LVEF < 30%
11. Severe pulmonary hypertension with pulmonary systolic pressure greater than two-thirds of systemic pressure
12. Hemodynamic instability requiring inotropic drug therapy within the past 14 days
13. Untreated clinically significant coronary artery disease requiring revascularization
14. Presence of significant aortic disease such as atheroma, thrombus, or aneurysm which, in the opinion of the investigator, precludes safe implant delivery
15. Blood dyscrasias defined as: acute leukopenia, acute anemia, acute thrombocytopenia, history of bleeding diathesis or coagulopathy
16. Patient ineligible for or refuses blood transfusions
17. Unfavorable peripheral vascular anatomy or disease (e.g. severe obstructive calcification, severe tortuosity or vessels < 6 mm) that would preclude passage of catheters from the femoral arterial access to the aorta as evidenced by peripheral MSCT
18. Active peptic ulcer or gastrointestinal bleeding within the past 90 days*
19. Symptoms of carotid or vertebral artery disease (e.g. stroke or transient ischemic attack) within past 6 month, or treatment of carotid stenosis within past two months*
20. Renal insufficiency as demonstrated by a serum creatinine > 2.5 mg/dL or end stage renal disease requiring chronic dialysis
21. Active infection requiring ongoing treatment
22. Need for emergent surgery or intervention other than the investigational procedure
23. Any therapeutic invasive cardiac procedure performed or planned to perform within 30 days of the index procedure except for PCI which is within 7 days of the index procedure*
24. Hypersensitivity or contraindication to procedural medication and device materials (e.g. titanium, nickel, pork) which cannot be adequately pre-medicated
25. Life expectancy < 1 year due to non-cardiac co-morbid conditions
26. Currently participating in any investigational drug or device studies that may confound the results of this study
27. History of any cognitive or mental health status that would interfere with study participation * At the time of procedure, if a subject's medical status has changed since enrollment, the subject shall be re-evaluated for eligibility.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Mortality at 30 days | 30 days
  The primary safety endpoint is all-cause mortality at 30 days

SECONDARY OUTCOMES:
Secondary Performance Endpoint 1: Procedural Device Performance | 1 day
  The secondary performance endpoint is Device Success defined as:
  * Absence of procedural mortality AND
  * Correct positioning of a single Valve into the proper anatomical location AND
  * Intended performance of the Valve (no severe prosthesis-patient mismatch and clinically acceptable gradient) AND no moderate or severe aortic valve regurgitation)
Secondary Performance Endpoint 2: Post-procedural Valve Performance (Aortic Valve Effective Orifice Area) | 1 week, 1, 6, 12, 24, 36, 48 and 60 months
  Aortic valve effective orifice area (EOA) will be evaluated with echocardiograms
Secondary Performance Endpoint 2: Post-procedural Valve Performance (Severity of Aortic Valve Regurgitation) | 1 week, 1, 6, 12, 24, 36, 48 and 60 months
  Severity of aortic valve regurgitation (AR) will be evaluated with echocardiograms
Secondary Performance Endpoint 2: Post-procedural Valve Performance (Aortic Valve Gradient) | 1 week, 1, 6, 12, 24, 36, 48 and 60 months
  Aortic valve gradient will be evaluated with echocardiograms
Secondary Safety Endpoint 3: Adverse Events | throughout the 5 year follow up period
  All adverse events will be assessed throughout the 5 year follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodés-Cabau, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval; Harindra Wijeysundera, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodes-Cabau J, Williams MR, Wijeysundera HC, Kereiakes DJ, Paradis JM, Staniloae C, Saric M, Radhakrishnan S, Wilson RF, Kubo SH. Transcatheter Aortic Valve Replacement With the HLT Meridian Valve. Circ Cardiovasc Interv. 2019 Aug;12(8):e008053. doi: 10.1161/CIRCINTERVENTIONS.119.008053. Epub 2019 Jul 31. PMID 31362540